CLINICAL TRIAL: NCT06813144
Title: Evaluation of the Effectiveness of Respiratory Muscle Training with a Mobile Application in the Early Postoperative Period After Lobectomy
Brief Title: Effectiveness of Respiratory Muscle Training with a Mobile Application After Lobectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Funda Sirakaya, PHD student, physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-30603717-050.04-2400055696
Record Dates: First submitted 2025-01-22; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Video Assisted Thoracic Surgery (VATS); Thoracic Surgery; Respiratory Muscle; Lung Cancer (NSCLC)
Keywords: lung cancer; vats; inspiratory muscle training
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind (participant and statistician)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Classic IMT (Active Comparator): Individuals who are between the ages of 18-65 and lung cancer patient, underwent lobectomy with video-assisted thoracic surgery.
  The group will receive standard postoperative physiotherapy and rehabilitation as well as classical inspiratory muscle strength training with the noninvasive Powerbreath Medic Plus device (POWERbreathe International Ltd., Warwickshire, England). Training will start with 40 percent of the initial MIP level and progress will be planned according to Modified Borg between 3-4. It will be repeated twice a day for 3 times 10 minutes. Training will start on the 1st postoperative day after the participants are transferred to the ward and they will be asked to continue at home. The progress plan will be adjusted by talking to the patient on the phone every 2 days after discharge.
  Interventions: Other: inspiratory muscle exercise
- IMT with mobile application (Experimental): Individuals who are between the ages of 18-65 and lung cancer patient, underwent lobectomy with video-assisted thoracic surgery.
  The group will receive standard postoperative physiotherapy and rehabilitation as well as inspiratory muscle training with the smart adapter support (POWERbreathe International Ltd., Warwickshire, England). Training will start with 40 percent of the initial MIP level and progress will be planned according to Modified Borg between 3-4. It will be repeated twice a day for 3 times 10 minutes. Training will start on the 1st postoperative day after the participants are transferred to the ward and they will be asked to continue at home. The progress plan will be adjusted by talking to the patient on the phone every 2 days after discharge.
  Interventions: Other: inspiratory muscle exercise
- control group (No Intervention): Individuals who are between the ages of 18-65 and lung cancer patient, underwent lobectomy with video-assisted thoracic surgery.
  This group will receive only standard physiotherapy and rehabilitation: respiratory exercises (thoracic expansion exercises, diaphragmatic breathing, incentive spirometry), mobilization and cough/huffing training. Participants will be advised to continue these exercises regularly at home.

INTERVENTIONS:
Other: inspiratory muscle exercise — Inspiratory muscle training will be given with or without smart adaptor.
  Arms: Classic IMT; IMT with mobile application

SUMMARY:
It has been observed that there are negative effects on respiratory muscle strength following lobectomy. This has led to the necessity of respiratory muscle training to mitigate these adverse effects. Most studies conducted so far focus on the late postoperative period, and there are only a few studies evaluating the effectiveness of early postoperative inspiratory muscle training (IMT). It is believed that this method could be useful for facilitating patient follow-up and increasing patient motivation through visual feedback.

DETAILED DESCRIPTION:
It has been observed that there are negative effects on respiratory muscle strength following lobectomy. This has led to the necessity of respiratory muscle training to mitigate these adverse effects. Most studies conducted so far focus on the late postoperative period, and there are only a few studies evaluating the effectiveness of early postoperative inspiratory muscle training (IMT). Additionally, there is currently no study assessing the effectiveness of IMT using a smart adapter in patients who have undergone lobectomy. It is believed that this method could be useful for facilitating patient follow-up and increasing patient motivation through visual feedback. The aim of this study is to examine the changes in respiratory muscle strength and exercise capacity in patients after lobectomy via VATS, comparing classical IMT, mobile application-supported IMT, and a control group that does not receive IMT.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being clinically stable,
* Being a lung cancer patient with a planned lobectomy with VATS,
* Being between the ages of 18-65,
* Being able to cooperate with the tests to be performed.

Exclusion criteria:

* Having any orthopedic or neurological problem that prevents walking,
* Having undergone any surgery related to the thoracic wall,
* Having diseases that will affect respiratory parameters such as severe heart failure, severe chronic obstructive pulmonary disease (COPD).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Inspiratory muscle strength | Measurements will be performed before surgery (the day before surgery), at discharge and during the follow-up period after surgery (10-15 days after discharge).
  Respiratory muscle strength will measure by measuring mouth pressure and using maximal inspiratory pressure (MIP) values.
Expiratory muscle strength | Measurements will be performed before surgery (the day before surgery), at discharge and during the follow-up period after surgery (10-15 days after discharge).
  Respiratory muscle strength will measure by measuring mouth pressure and using maximal expiratory pressure (MEP) values.

SECONDARY OUTCOMES:
Functional exercise capacity | Evaluations will be made before surgery (the day before surgery) and during the follow-up period (10-15 days after discharge).
  6-minute walk test (6MWT) will be used to evaluate functional exercise capacity.
Postoperative Pulmonary Complications | Postoperative first-fifth days.
  Postoperative pulmonary complications will be evaulate by Melbourne Group Scale. If more than 4 parameters are positive, it will be considered as having postoperative pulmonary complication.
Exercise Motivation | The evaluation will be made during the control period (10-15 days after discharge).
  Exercise Motivation Attitude Scale will be used. This scale consists of 3 sub-dimensions (negative attitude and thought/positive view and health/physical appearance and health).
Dyspnea Level | An evaluation will be made in the preoperative (the day before surgery) and control period (10-15 days after discharge).
  Modified Borg Scale will be used to evaluate dyspnea.
Quality of Life | The evaluation will be made during the preoerative (the day before surgery) and control (10-15 days after discharge) period.
  SF-12 Quality of Life Scale will be used to assess quality of life.
Physical Performance | Evaluations will be made in the preoperative (the day before surgery) and control (10-15 days after discharge) periods.
  The Short Physical Performance Battery, a frequently used test in cardiovascular and pulmonary diseases, will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, Professorr, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided